CLINICAL TRIAL: NCT06859827
Title: The Role of Cardiac MRI Feature Tracking in Assessment of Hypertrophic Cardiomyopathy and Athlete's Heart.
Brief Title: Role of CMR-FT in Assessment of HCM and Athlete's Heart.
Status: Active, not recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Abdelrahman Abdelmageed Ragab, Assistant lecturer diagnostic and interventional radiology, Sohag University
Other Study IDs: Soh-Med-25-2--MD
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Hypertrophic Cardiomyopathies; Athlete Heart
Keywords: Cardiac MRI feature tracking; Hypertrophic cardiomyopathy; Athlete's heart
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- hypertrophic cardiomyopathy patient: patient with hypertrophic cardiomyopathy
- Athlete's: Athlete's with thick myocardium

SUMMARY:
Using cardiac MRI feature tracking to asses myocardial motion differences in athlete's heart and discovered hypertrophic cardiomyopathy patients to increase diagnostic accuracy of hypertrophic cardiomyopathy.

DETAILED DESCRIPTION:
Cardiac MRI is the gold standard for assessing cardiac function without significant limitations of anatomical restrictions. CMR-FT helps in assessment of myocardial deformation on routinely obtained by steady state free precision (SSFP) cine images. CMR-FT is used in cardiac research and became common in clinical practice. It has been used in assessment of wide spectrum of cardiac diseases and provides for comprehensive and reliable assessments of heart function.

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected to be hypertrophic cardiomyopathy by echocardiography..
* Athletes and heavy workers,, healthy volunteers also included.

Exclusion Criteria:

* Patients with absolute or relative contraindications to magnetic resonance imaging (e.g intra-ocular metallic foreign body, claustrophobia, etc) or contra-indication to MRI contrast medium.
* Clinical morbidities with absolute contraindication to anesthesia during the examination in un-cooperative patients where sedation is required.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Any age between 20 and 50 years either male or female with minor complains and suspected by Echo to be hypertrophic cardiomyopathy, athlete's exhibiting no symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Use of cardiac MRI feature tracking in detection of myocardial deformation abnormalities and diagnostic confirmation and detection of hypertrophic cardiomyopathy. | 6months to 12 months
  The main goal of the study is evaluating the role of Cardiac magnetic resonance feature tracking analysis in detection of myocardial deformation abnormalities in cases of hypertrophic cardio myopathy and compare it with physiological hypertrophy in athletes.
  Identification of strain patterns in hypertrophic cardiomyopathy.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospital, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided